CLINICAL TRIAL: NCT03374345
Title: Efficacy and Safety of Sipjeondaebo-tang on Korean Patients With Cold Hypersensitivity in the Hands and Feet (SDT)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gachon University Gil Oriental Medical Hospital (Other)
Collaborators: Kyunghee University Medical Center (Other); Kyung Hee University Hospital at Gangdong (Other); Semyung University Affiliated Oriental Medical Hospital (Other); Sangji University Oriental Medical Hospital (Unknown)
Responsible Party: Principal Investigator, Chan-Yong Jeon, Principle Investigator, Gachon University Gil Oriental Medical Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISEE_2017_SDT
Record Dates: First submitted 2017-11-27; First posted 2017-12-15 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Cold Hypersensitivity
Keywords: Cold Hypersensitivity; Korean medicine; Sipjeondaebo-tang; Cold intolerance
MeSH Terms: conditions — Cold Hypersensitivity | interventions — juzentaihoto

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDT group (Experimental): 3g, three times a day, each taken before or between meals Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Interventions: Drug: Sipjeondaebo-tang Granule
- Placebo group (Placebo Comparator): 3g, three times a day, each taken before or between meals Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sipjeondaebo-tang Granule — 3g, three times a day, each taken before or between meals Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Other Names: Deciten Granule
  Arms: SDT group
Drug: Placebo — 3g, three times a day, each taken before or between meals Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Arms: Placebo group

SUMMARY:
Gachon University, Gil Oriental Medicine Center

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 19 to 59 years have a complaint of CHH.
* Patients must include at least one or more of the following symptoms:
* Those who have the symptoms of CHH in normal temperature which most individuals feel no cold;
* Those who have the symptoms of extremely cold hands in cold temperature exposure;
* Those who are on the return to a warmer environment, the symptoms of cold hands is not completely rewarmed;
* Those who have 4 cm or greater of VAS CHH score;
* A thermal differences between the palm (PC8) and the upper arm (LU4) may be higher than 0.3℃;
* Those who can comply with all study-related procedures, medications, and evaluations;
* Given a written informed consent form.

Exclusion Criteria:

* Patients with calcium antagonists or beta-blockers with the purpose of treating CHH;
* Those who have one or more finger gangrene or ulceration;
* Those who are diagnosed by hypothyroidism or currently medicated to thyroid drugs;
* Those who are diagnosed by autoimmune disease or have a positive ANA test result;
* Those who are diagnosed by carpal tunnel syndrome or have a positive Tinel and Phalen's tests;
* Those who are diagnosed with cervical disc herniation or (malignant) tumor disease;
* Those who are diagnosed with diabetes;
* Those who are currently medicated to drugs that may affect to CHH symptoms, such as anticoagulants etc;
* Those who have moderate level of liver dysfunction (each of AST, ALT greater than 100 IU/L) or kidney dysfunction (Cr 2.0mg/dL);
* Those who do not (cannot) abide by treatment and follow up due to the mental illness such as behavior disorder, depression, anxiety neurosis, schizophrenia, or serious mental illness;
* Those who are Diagnosed with moderate anemia and hematologic disorders (adult non-pregnant women hemoglobin (Hgb) level less than 7g/dL, hematocrit (Hct) level less than 26%, white blood cell (WBC) level greater than 11,000/mm3); Those whose systolic blood pressure (SBP) 180mmHg or diastolic blood pressure (DBP) is greater than 100 mmHg based on average value of at least 2 measurements;
* Those who are suspected arrhythmia that showing up on ECG, or diagnosed by heart diseases, such as, ischemic heart disease and so on;
* Those who are addicted to alcohol or drugs;
* Those who are pregnant (positive urine-HCG) or lactating or have the chances of pregnancy;
* Those who are diagnosed with malignant tumor
* Those who are currently participated in other clinical trials;
* Those who are able to understand and speak Korean;
* Those who are judged to be inappropriate for the clinical study by the researchers.

Ages: 19 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in visual analogue scale(VAS) | At baseline, week 4, 8, 12
  The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels.

SECONDARY OUTCOMES:
Changes from baseline in body temperature | At baseline, week 4, 8, 12
  Changes from baseline in body temperature
Changes from baseline in WHO Quality of Life-BREF | At baseline, week 4, 8, 12
  It is a international cross-culturally comparable quality of life assessment instrument. The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. There are also two items that are examined separately: Q1 asks about an individuals overall perception of QoL and Q2 asks about an individuals overall perception of their health. The four domain scores denote an individuals perception of QoL in each particular domain. Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life). The mean score of items within each domain is used to calculate the domain score. Meanscores are then multiplied by 4 in order to make domain scores comparable with the scores used in the WHOQOL-100.
Changes from baseline in blood pressure | up to 12 weeks
  assess for monitoring patient safety
Changes from baseline in Pulse rate | up to 12 weeks
  assess for monitoring patient safety
Levels of AST | At screening visit, week 8
  liver function test for monitoring patient safety(IU/L)
Levels of ALT | At screening visit, week 8
  liver function test for monitoring patient safety(IU/L)
Levels of r-GTP | At screening visit, week 8
  liver function test for monitoring patient safety(IU/L)
Levels of BUN | At screening visit, week 8
  Kidney function test for monitoring patient safety(mmol/L)
Levels of Cr | At screening visit, week 8
  Kidney function test for monitoring patient safety(mmol/L)
complete blood count | At screening visit, week 8
Adverse event | At week 4, 8, 12

OTHER OUTCOMES:
Pattern Identification Questionnaire | At screening visit
  This tool is a traditional medicine researcher self-developed questionnaire of screening for patients with Cold Hypersensitivity in the Hands and feet In this trial, we will assess the validity of the tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ko Y, Sun SH, Han IS, Go HY, Kim TH, Lee JM, Jang JB, Park KS, Song YK, Lee KY, Jeon CY, Ko SG. The efficacy and safety of Sipjeondaebo-tang in Korean patients with cold hypersensitivity in the hands and feet: a protocol for a pilot, randomized, double-blind, placebo-controlled, parallel-group clinical trial. Trials. 2019 Apr 15;20(1):217. doi: 10.1186/s13063-019-3286-7. PMID 30987667